CLINICAL TRIAL: NCT03023241
Title: Diagnosis of Bladder Pain Syndrome / Interstitial Cystitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cantonal Hospital, Frauenfeld (Other)
Responsible Party: Principal Investigator, Prof. Dr. Volker Viereck, Prof. Dr. med., Cantonal Hospital, Frauenfeld
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 9900.013 BPS/IC study; KEKTGOV2010/01 (Other: Canton Thurgau Ethics Commission)
Record Dates: First submitted 2017-01-13; First posted 2017-01-18 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Bladder Pain Syndrome; Interstitial Cystitis; Overactive Bladder
Keywords: BPS/IC; OAB
MeSH Terms: conditions — Cystitis, Interstitial; Urinary Bladder, Overactive | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- all study patients (Experimental): Same intervention for all subjects: anamnesis, questionnaires and biological samples (bladder biopsy, bladder washing, blood and urine) are collected at one single visit.
  Interventions: Procedure: biopsy

INTERVENTIONS:
Procedure: biopsy — cold cup bladder biopsies and bladder washings under anesthesia, blood and urine collection

SUMMARY:
To identify new, simple and reliable biomarkers for bladder pain syndrome/interstitial cystitis (BPS/IC) for diagnosis of this disease.

DETAILED DESCRIPTION:
Collection and analyses of bladder biopsies, bladder washings, blood and urine samples of patients with bladder pain syndrome/interstitial cystitis (BPS/IC), overactive bladder syndrome (OAB) and bladder-healthy controls. Analyses include ELISA, RT-qPCR, DNA sequencing, and immunohistochemistry techniques. Differences between patient groups are statistically evaluated.

ELIGIBILITY:
Inclusion Criteria:

* patient with diagnosed BPS/IC, OAB or healthy controls
* included healthy controls must have another pelvic surgery planned (e.g. hysterectomy)
* being able to act and judge

Exclusion Criteria:

* unstable endocrinological situation
* severe illness

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2004-12; Primary Completion 2020-12 (Actual); Study Completion 2021-07 (Actual)

PRIMARY OUTCOMES:
Identification of new diagnostic markers for BPS/IC | 2 days

SECONDARY OUTCOMES:
Identification of molecular details that lead to BPS/IC (pathogenesis). | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Volker Viereck, Prof. Dr., Principal Investigator — Cantonal Hospital Frauenfeld, Switzerland
Locations (1):
- Cantonal Hospital Frauenfeld, Frauenfeld, Thurgau, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gamper M, Viereck V, Geissbuhler V, Eberhard J, Binder J, Moll C, Rehrauer H, Moser R. Gene expression profile of bladder tissue of patients with ulcerative interstitial cystitis. BMC Genomics. 2009 Apr 28;10:199. doi: 10.1186/1471-2164-10-199. PMID 19400928
- [Result] Gamper M, Viereck V, Eberhard J, Binder J, Moll C, Welter J, Moser R. Local immune response in bladder pain syndrome/interstitial cystitis ESSIC type 3C. Int Urogynecol J. 2013 Dec;24(12):2049-57. doi: 10.1007/s00192-013-2112-0. Epub 2013 May 14. PMID 23670165
- [Result] Gamper M, Regauer S, Welter J, Eberhard J, Viereck V. Are mast cells still good biomarkers for bladder pain syndrome/interstitial cystitis? J Urol. 2015 Jun;193(6):1994-2000. doi: 10.1016/j.juro.2015.01.036. Epub 2015 Jan 14. PMID 25596361
- [Result] Gamper M, Moser R, Viereck V. Have we been led astray by the NGF biomarker data? Neurourol Urodyn. 2017 Jan;36(1):203-204. doi: 10.1002/nau.22882. Epub 2015 Sep 18. No abstract available. PMID 26384156
- [Result] Regauer S, Gamper M, Fehr MK, Viereck V. Sensory Hyperinnervation Distinguishes Bladder Pain Syndrome/Interstitial Cystitis from Overactive Bladder Syndrome. J Urol. 2017 Jan;197(1):159-166. doi: 10.1016/j.juro.2016.06.089. Epub 2016 Jul 1. PMID 27378135